CLINICAL TRIAL: NCT07195240
Title: The Effect of Lemongrass on Aerobic Performance and Sexual Wellbeing Following High-Intensity Interval Training Training in Middle Aged Males
Brief Title: The Effect of Lemongrass on Aerobic Performance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Mibelle Group Biochemistry (Industry)
Responsible Party: Principal Investigator, Glyn Howatson, Professor, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 10394
Record Dates: First submitted 2025-09-05; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Sexual Wellness; Aerobic Capacity; Exercise Efficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active: Lemongrass Extract (Experimental): Tablet containing 200mg Lemongrass extract (Mibelle).
  Interventions: Dietary Supplement: Active: Lemongrass
- Control: Placebo (Experimental): Tablet containing microcrystalline cellulose.
  Interventions: Dietary Supplement: Control: Placebo

INTERVENTIONS:
Dietary Supplement: Active: Lemongrass — 200mg of lemongrass extract
  Arms: Active: Lemongrass Extract
Dietary Supplement: Control: Placebo — microcrystalline cellulose
  Arms: Control: Placebo

SUMMARY:
The goal of this experimental study is to examine the influence of Lemongrass extract on aerobic training parameters following a 6-week training programme in middle-aged males. A secondary aim will be to explore the influence on sexual wellness. Participants will attend 23 visits to the laboratory involving:

* fitness testing (some to exhaustion).
* blood sampling (capillary and venous samples).
* a supervised 6 week high-intensity interval training (HIIT) programme.
* consuming either the lemongrass extract or placebo in the form of tablets, once a day during the 6 week training.

DETAILED DESCRIPTION:
The study is a randomised, parallel (two groups, lemongrass versus placebo), double-blind, placebo-controlled design in middle-aged males (40-60 years).

Visit 1: Pre-screening Participants will receive information on the study, be assessed for contraindications, be familiarised with the requirements for participation, and provide written informed consent.

Visit 2: Familiarisation with the dependent measures Study staff will review physical activity questionnaires, and if eligibility criteria are met, participants will enter the trial. Participants will refrain from physical activity and alcohol consumption for 24 hours, and caffeine for 12 hours before each visit. Next, participants will be familiarised with the equipment to be used during the study.

Following a resting capillary blood lactate sample, participants will perform an exercise session on a cycle ergometer, beginning with a 5-minute warm-up at a self-paced intensity equating to approximately 10 on the 6-20 Rating of Perceived Exertion (RPE) scale.

The session will then start with the participant cycling at 50 watts (W) for 4 minutes, with an increase of 30 W every 4 minutes, while blood lactate is taken and heart rate recorded in the last 30 seconds of each stage. Once blood lactate has reached the second inflection point, the test will be terminated. Throughout the exercise session, expired air will be measured using online gas analysis.

Visit 3: Baseline measures Participants will report to the laboratory in a fed and hydrated state, having avoided strenuous activity for 24 hours, where baseline measurements of all dependent variables will be taken. Participants will complete a food diary for the 24-hour period prior to testing. The diary will be analysed using dietary analysis software, and participants will be instructed to replicate all food and fluid intake prior to the follow-up testing visit.

Upon arrival, a venous blood sample will be collected via the antecubital fossa, which will be frozen and stored for subsequent analysis of exercise-affected metabolites. Participants will then complete a sexual wellbeing questionnaire.

Following this, participants will repeat the submaximal protocol described in Visit 2. After a rest period of 10 minutes, participants will complete a graded exercise protocol to determine peak oxygen uptake (VO₂peak). The test will start at the intensity immediately below the second inflection point identified on the lactate profile. The intensity will increase by 30 W each minute until VO₂peak is achieved, which will be confirmed when at least one of the following criteria is met:

* A plateau in VO₂ despite an increase in workload;
* A respiratory exchange ratio (RER) higher than 1.15;
* Peak heart rate at least equal to 90% of the age-predicted maximum;
* RPE greater than 18;
* Blood lactate concentration greater than 8 millimoles per litre (mmol·L-¹).

Maximum aerobic power will be defined as the final completed work rate. This will be used for subsequent training prescription (125% of maximal aerobic power [Pmax]).

Upon completion, participants will be supplied with their assigned product (lemongrass or placebo). They will consume one capsule daily, taken with the main meal prior to training sessions, with this timing repeated on non-training days.

6-Week Training Intervention (Visits 4-22) Participants will be required to attend three training sessions per week for a total duration of six weeks. Participants will complete a series of 30-second efforts at 125% of maximum Pmax (determined during the VO₂peak test), followed by 2 minutes of recovery.

In weeks 1-5, participants will complete 6, 7, 8, 9, and 10 intervals per session, respectively.

In week 6, participants will complete 8 intervals per session (to replicate a taper).

Each session will begin with a 5-minute, self-paced warm-up. Participants will maintain their habitual physical activity pattern between visits. Any exercise outside of the study will be recorded.

Visit 23: Post-training intervention testing Participants will repeat Visit 3 and complete all dependent measures within 48 hours of the final training session.

A follow-up communication via telephone will be conducted within 7 days of completion of the final session to ensure there are no adverse effects from participation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 and ≤ 60 years.
* Body Mass Index (BMI) ≥ 19 and ≤ 35 kg/m2.
* Willingness and ability to comply with the protocol in the opinion of the Investigator.
* Judged by the Investigator to be in good health as assessed by a health screening questionnaire.
* Currently identifies as the same biological sex as at birth.
* Currently deemed to be sedentary or relatively inactive (less than 150 minutes of moderate physical activity per week).
* Have a blood pressure < 140/90 mmHg.

Exclusion Criteria:

* A history of heart disease.
* Any disease that might interfere with the absorption of nutrients (e.g. Chron's disease, celiac disease).
* Recent musculoskeletal or soft tissue injury (within the last 3 months).
* The habitual use of medication that is antihypertensive or antidiabetic medication or might inhibit the ability to complete the study participation.
* Alcohol Intake of greater than 21 units per week.
* A change in bodyweight of more than 3kg within the month preceding the study.
* Currently following a weight-loss or weight-gain programme.
* Any known bleeding disorder or reaction to withdrawal of blood samples

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Aerobic Capacity | This measure will assessed and measured twice: Baseline assessment: Visit 3 (Week 1, prior to the intervention). Post-intervention assessment: Visit 23 (Week 8, within 48 hours after the final training session).
  To determine the effect of the intervention vs placebo on marker of aerobic capacity (VO2peak). It will be assessed using breath-by-breath gas analysis during a graded exercise protocol on a static bike. The test will start at the intensity immediately below the second inflection point identified on the lactate profile (conducted in visit 2). The intensity will increase by 30 w each minute until VO2peak which will be confirmed when at least one of the following criteria (according to CASES) are met: (1) a plateau in VO2 despite an increase in workload; (2) a respiratory exchange ratio (RER) higher than 1.15; (3) peak heart rate at least equal to 90% of the age-predicted maximum and/or (4) RPE of >18; (5) a blood lactate concentration of > 8mMol/L. Maximum aerobic power will be defined as the final completed work rate. This will be used for subsequent training prescription (125% of maximal aerobic power [Pmax]).
Aerobic Performance (blood lactate) | This measure will be assessed three times. Familiarisation and lactate profiling: Visit 2 (Week 0). Baseline assessment: Visit 3 (Week 1, prior to the intervention), Post-intervention assessment: Visit 23 (Week 8, within 48 hrs after the final training).
  To determine the effect of intervention vs placebo on secondary markers of maximal aerobic performance (blood lactate). A total of 14 (more if the submaximal exercise test progresses beyond 4 stages) capillary samples will be collected for each participant during the submaximal and graded exercise tests. This will be pre-exercise, then in the final minute of each ramped stage during the submaximal test. A final lactate sample will be collected upon completion of the VO2peak test. These samples will be analysed for lactate concentration immediately using a Biosen C-line analyser before being disposed of.
Aerobic Performance (heart rate) | This measure will be assessed three times. Familiarisation and lactate profiling: Visit 2 (Week 0). Baseline assessment: Visit 3 (Week 1, prior to the intervention), Post-intervention assessment: Visit 23 (Week 8, within 48 hrs after the final training).
  To determine the effect, if any, of intervention vs placebo on secondary markers of maximal aerobic performance (heart rate). Heart rate will be continuously monitored using a chest strap (Polar monitor) throughout the various exercise protocols (lactate profiling in visit 2 and 3, and the graded exercise task in visit 3 and 23).

SECONDARY OUTCOMES:
Sexual Wellness | This measure will assessed and measured twice: Baseline assessment: Visit 3 (Week 1, prior to the intervention). Post-intervention assessment: Visit 23 (Week 8, within 48 hours after the final training session).
  To determine, if any, changes in sexual wellbeing resulting from the intervention. Sexual wellbeing will be defined using a sexual function questionnaire (DISF-SR). Derogatis interview for sexual functioning-self report, set of 21 questions, split into four domains: sexual cognition/ fantasy, sexual arousal, sexual behaviour/ experiences and orgasm.
Serum | This measure will assessed and measured twice: Baseline assessment: Visit 3 (Week 1, prior to the intervention). Post-intervention assessment: Visit 23 (Week 8, within 48 hours after the final training session).
  A total of 2 venous blood samples will be taken during visit 3 and visit 23, and serum will later be analysed for biomarkers associated with exercise metabolism to assess what effect, if any, the intervention has had on metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria Univeristy
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No